CLINICAL TRIAL: NCT02412709
Title: ECG Device for Long QT Syndrome Screening in Newborns
Brief Title: Long QT Syndrome Screening in Newborns
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: QT Medical, Inc. (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Ruey-Kang Chang, Chief Executive Officer, QT Medical, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 30147-01
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Long QT Syndrome
Keywords: Long QT Syndrome; LQTS; genetic testing; ECG; saliva testing
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Performing ECG (PPE) (Experimental): Parent Performing ECG (PPE) Group--When the baby is 2 weeks old, research staff will contact interested parents to schedule a home visit. During the visit, a research assistant will provide the parents with a kit that includes the QTScreen system and instructions. The parents will perform an ECG on their child using the QTScreen and instructions. If after attempting the ECG on their own parents encounter problems, parents can ask the research assistant for assistance.
  Interventions: Device: QTScreen ECG Recorder
- Staff Performing ECG (SPE) (Active Comparator): Staff Performing ECG (SPE) Group--When the baby is 2-4 weeks of age, research staff will contact the family to schedule a home visit. The QTScreen test will be done by a research assistant.
  Interventions: Device: QTScreen ECG Recorder

INTERVENTIONS:
Device: QTScreen ECG Recorder — Subjects will be randomly assigned to the: Parents Performing ECG (PPE) group or Staff Performing ECG (SPE) group. This will assess whether parents are able to use QTScreen on babies at home.

SUMMARY:
The purpose of this project is to test a new, very compact, 12-lead ECG device as a way to detect long QT syndrome (LQTS) in infants. The device -- called QTScreen -- was developed in Phase I of this project.

In Phase II, the goals are to test the capacity of the device for LQTS screening in newborns and to obtain prevalence data on LQTS in California.

The 4 main objectives are:

1. To validate the capacity of QTScreen for LQTS screening in newborns.
2. To determine the extent to which parents are able to use QTScreen on their babies at home.
3. To survey end-user experience and opinions.
4. To estimate the LQTS prevalence in California.

DETAILED DESCRIPTION:
Long QT syndrome (LQTS) is a genetic disorder characterized by a prolonged QT interval on the ECG and occurrence of syncope, ventricular arrhythmias, and sudden death. LQTS is a major cause of sudden death in infants, children, and young adults. Treatment by β-blockers and/or placement of an implantable cardioverter defibrillator (ICD) are effective in preventing sudden death, if the diagnosis of LQTS is made early.

The efficacy of ECG screening of newborns for LQTS has been demonstrated in Italy. Furthermore, within the national healthcare system in Italy, universal ECG screening in newborns (<30 days old) is cost-effective. The U.S. debate for universal LQTS screening started in the mid-2000's. In a 2007survey completed by North American pediatric cardiologists, 27% favored optional ECG screening of newborns, whereas 11% supported mandatory screening (363 responses, 35% response rate). There may be stronger support for universal screening, now that more data are available.

Obtaining a good standard 12-lead EKG on a neonate in the clinic is difficult and time consuming. If an ECG device for newborn screening were readily available, reliable, easy to use, and cost-effective, then universal screening of all 4 million newborns in the U.S. each year would identify 2,000 infants with LQTS who are at risk for sudden death, assuming the prevalence is the same as in Italy. Perhaps more than 300 deaths per year from SIDS could be prevented, as well as many more sudden deaths in children, adolescents, and young adults.

During Phase I of this project, a new device was developed to meet this clinical need (called QTScreen). In Phase II, the aim is to test the capacity of QTScreen for LQTS screening in newborns and the feasibility of home screening by parents in an ethnically diverse population of Northern and Southern California. The results of this clinical trial may validate the device as a screening tool for LQTS, and also provide important scientific data for supporting newborn screening for LQTS in the U.S.

The 4 main objectives are:

1. To validate the capacity of QTScreen for LQTS screening in newborns. This will be a clinical trial on 4,000 newborns, conducted at the Los Angeles Biomedical Research Institute (LABioMed).
2. To determine the extent to which parents are able to use QTScreen on their babies at home.
3. To survey end-user experience and opinions. The target users of QTScreen are parents. Participating parents will be asked to complete a survey, to obtain data for further development of the device.
4. To estimate the LQTS prevalence in California. To date, the only population-based estimate of LQTS prevalence is 1 in 2,000 in Italy. In a recent study in Japan, 4,285 1-month-old infants had ECG screening. The LQTS prevalence was not reported, because only 10% of subjects with QTc values >450 msec had gene testing. There has been no population-based study of LQTS in the US. In a study of 707 children with hearing loss in California, 2 subjects had potassium voltage-gated channel KQT-like subfamily member 1 (KCNQ1 potassium channel) mutations, truncation or splicing. This trial will provide data on the LQTS prevalence in California.

Study Sites:

Study procedures will be conducted at subjects' homes. Subjects will be recruited from LA BioMed at Harbor-UCLA Medical Center, Providence Little Company of Mary Medical Center-Torrance, Santa Clara Valley Medical Center, and St. Francis Medical Center. Approval from each of the recruitment sites will be obtained prior to commencing recruitment.

Consent:

Consent will be sought from one parent only. Parents will be given the opportunity to thoroughly read the consent form and to ask questions.

Risk/Benefit:

ECG is a routine test performed on infants, children and adults every day in the hospital for many years with no problems or adverse events. The QTScreen system used in this study is a simplified way of performing an ECG test on infants. Some subjects may undergo genetic testing as part of this research and there are some risks associated with genetic testing, such as emotional and confidentiality.

There is a very small risk of infection or rash related to the procedure involved in ECG testing. The subject may feel some discomfort from the sticky patches placed on and removed from his/her chest. Discomfort will be minimized by using an adhesive remover wipe which is commercially available and used by hospitals. Although infection is very unlikely to occur, rules and procedures of the nursery and clinic will be followed. This includes cleaning the ECG equipment and sanitizing it using a disinfecting wipe before and after each use to prevent infection.

The effects of drawing blood are usually pain, bleeding and/or a bruise where the needle is inserted. Occasionally the area around the vein may swell. Serious complications such as a blood clot or infection may occur but these are rare. Some people feel faint when having blood drawn. Necessary precautions, such as gloves and proper sterilization, will be taken to minimize pain and infection. A small amount of local anesthetic cream may be placed on the child's forearm.

Appropriate precautions will be used to minimize the risks associated with this project and feel that in general the risks associated with this project are low.

The information gained from this study will help to find ways to possibly simplify the ECG test. This research study may also lead to a better understanding of LQTS which can provide important insight for future treatments and research. Therefore the general feeling is that the benefits of this project outweigh the risks.

ELIGIBILITY:
Inclusion Criteria:

1. Born at ≥36 weeks of gestation.
2. Birth weight 2.5-4.5 kg

Exclusion Criteria:

1. Babies that have been born with a heart disease.
2. Babies who have a skin condition, allergies, or chest deformities making ECG on the chest difficult or impossible.

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Determine LQTS risk via QTc Measurement and family/personal history | within 1-2 business days after QTScreen recording
  A standard 12-lead ECG will be printed from the QTScreen recording. Investigators will manually measure a corrected QT interval (QTc) from lead II, and examine any clinical ECG abnormalities. Subjects with a positive history, or subjects with a median QTc ≥450 ms on the first QTScreen will be categorized as Intermediate Risk and undergo a repeat QTScreen in 2-4 weeks (before 2 months of age).
Determine if parents are able to use QTScreen on babies at home | 18 to 24 months (within 6 months after the clinical trial is completed)
  Participants in the PPE group will be provided with the QTScreen recording device along with instructions for conducting an ECG on their baby. While conducting the ECG, a research assistant will access the parents' ability in properly conducting the ECG via a questionnaire.

SECONDARY OUTCOMES:
Follow-up for false negatives and survey end-user experience | at 1 year after LQTS screening
  A research assistant will conduct a follow-up of each subject when the subject turns 1 year of age. For subjects <1 year of age when the project ends, the family will be contacted at the end of the project period and when the subject turns 1 year. Parents will be inquired about: any diagnosis of LQTS, heart disease, fainting, seizures, or sudden death (SIDS) after the screening. If a subject had fainting or seizures but no subsequent cardiac evaluation, he/she will be scheduled for a repeat QTScreen. If a subject died of sudden unexplained death or SIDS, the parents will be offered ECG and genetic testing for LQTS. After the follow-up questions, parents will be surveyed on their experience with QTScreen.
Estimate the LQTS prevalence in California | 18 to 24 months (within 6 months after the clinical trial is completed)
  The large sample size and use of genetic conformation in this study provides a unique opportunity to evaluate the LQTS prevalence, as well as differences in certain ethnic groups, such as Latinos and White. The number of subjects with confirmed LQTS includes true positives, identified by positive QTScreen testing followed by gene testing, and false negatives identified by telephone follow up and subsequent confirmation. Prevalence data will be reported as the proportion of subjects with confirmed LQTS (and binomial exact 95% CI).

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Kang Chang, M.D., M.P.H., Principal Investigator — QT Medical, Inc.
Locations (3):
- United States (3):
  - St. Francis Medical Center, Lynwood, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Providence Little Company of Mary Medical Center-Torrance, Torrance, California

REFERENCES:
- [Background] Schwartz PJ, Stramba-Badiale M, Crotti L, Pedrazzini M, Besana A, Bosi G, Gabbarini F, Goulene K, Insolia R, Mannarino S, Mosca F, Nespoli L, Rimini A, Rosati E, Salice P, Spazzolini C. Prevalence of the congenital long-QT syndrome. Circulation. 2009 Nov 3;120(18):1761-7. doi: 10.1161/CIRCULATIONAHA.109.863209. Epub 2009 Oct 19. PMID 19841298
- [Background] Ackerman MJ, Siu BL, Sturner WQ, Tester DJ, Valdivia CR, Makielski JC, Towbin JA. Postmortem molecular analysis of SCN5A defects in sudden infant death syndrome. JAMA. 2001 Nov 14;286(18):2264-9. doi: 10.1001/jama.286.18.2264. PMID 11710892
- [Background] Tester DJ, Ackerman MJ. Sudden infant death syndrome: how significant are the cardiac channelopathies? Cardiovasc Res. 2005 Aug 15;67(3):388-96. doi: 10.1016/j.cardiores.2005.02.013. PMID 15913580
- [Background] Arnestad M, Crotti L, Rognum TO, Insolia R, Pedrazzini M, Ferrandi C, Vege A, Wang DW, Rhodes TE, George AL Jr, Schwartz PJ. Prevalence of long-QT syndrome gene variants in sudden infant death syndrome. Circulation. 2007 Jan 23;115(3):361-7. doi: 10.1161/CIRCULATIONAHA.106.658021. Epub 2007 Jan 8. PMID 17210839
- [Background] Weese-Mayer DE, Ackerman MJ, Marazita ML, Berry-Kravis EM. Sudden Infant Death Syndrome: review of implicated genetic factors. Am J Med Genet A. 2007 Apr 15;143A(8):771-88. doi: 10.1002/ajmg.a.31722. PMID 17340630
- [Background] Schwartz PJ, Crotti L. Can a message from the dead save lives? J Am Coll Cardiol. 2007 Jan 16;49(2):247-9. doi: 10.1016/j.jacc.2006.10.009. Epub 2006 Dec 29. No abstract available. PMID 17222737
- [Background] Gajewski KK, Saul JP. Sudden cardiac death in children and adolescents (excluding Sudden Infant Death Syndrome). Ann Pediatr Cardiol. 2010 Jul;3(2):107-12. doi: 10.4103/0974-2069.74035. PMID 21234187
- [Background] Van Hare GF, Perry J, Berul CI, Triedman JK. Cost effectiveness of neonatal ECG screening for the long QT syndrome. Eur Heart J. 2007 Jan;28(1):137; author reply137-9. doi: 10.1093/eurheartj/ehl414. Epub 2006 Dec 8. No abstract available. PMID 17158522
- [Background] van Langen IM, Wilde AA. Con: Newborn screening to prevent sudden cardiac death? Heart Rhythm. 2006 Nov;3(11):1356-9. doi: 10.1016/j.hrthm.2006.07.015. Epub 2006 Oct 11. No abstract available. PMID 17074645
- [Background] Chang RK, Rodriguez S, Gurvitz MZ. Electrocardiogram screening of infants for long QT syndrome: survey of pediatric cardiologists in North America. J Electrocardiol. 2010 Jan-Feb;43(1):4-7. doi: 10.1016/j.jelectrocard.2009.07.004. PMID 19665725
- [Background] Schwartz PJ. Pro: Newborn ECG screening to prevent sudden cardiac death. Heart Rhythm. 2006 Nov;3(11):1353-5. doi: 10.1016/j.hrthm.2006.07.016. Epub 2006 Oct 10. No abstract available. PMID 17074644
- [Background] Chang RK, Lan YT, Silka MJ, Morrow H, Kwong A, Smith-Lang J, Wallerstein R, Lin HJ. Genetic variants for long QT syndrome among infants and children from a statewide newborn hearing screening program cohort. J Pediatr. 2014 Mar;164(3):590-5.e1-3. doi: 10.1016/j.jpeds.2013.11.011. Epub 2013 Dec 31. PMID 24388587
- [Background] Schwartz PJ. The congenital long QT syndromes from genotype to phenotype: clinical implications. J Intern Med. 2006 Jan;259(1):39-47. doi: 10.1111/j.1365-2796.2005.01583.x. PMID 16336512
- [Background] Meyer JS, Mehdirad A, Salem BI, Kulikowska A, Kulikowski P. Sudden arrhythmia death syndrome: importance of the long QT syndrome. Am Fam Physician. 2003 Aug 1;68(3):483-8. PMID 12924831
- [Background] Tester DJ, Kopplin LJ, Creighton W, Burke AP, Ackerman MJ. Pathogenesis of unexplained drowning: new insights from a molecular autopsy. Mayo Clin Proc. 2005 May;80(5):596-600. doi: 10.4065/80.5.596. PMID 15887426
- [Background] Tester DJ, Ackerman MJ. Postmortem long QT syndrome genetic testing for sudden unexplained death in the young. J Am Coll Cardiol. 2007 Jan 16;49(2):240-6. doi: 10.1016/j.jacc.2006.10.010. Epub 2006 Dec 29. PMID 17222736
- [Background] Choi GR, Porter CB, Ackerman MJ. Sudden cardiac death and channelopathies: a review of implantable defibrillator therapy. Pediatr Clin North Am. 2004 Oct;51(5):1289-303. doi: 10.1016/j.pcl.2004.04.015. PMID 15331285
- [Background] Chatrath R, Bell CM, Ackerman MJ. Beta-blocker therapy failures in symptomatic probands with genotyped long-QT syndrome. Pediatr Cardiol. 2004 Sep-Oct;25(5):459-65. doi: 10.1007/s00246-003-0567-3. Epub 2004 Jul 30. PMID 15534720
- [Background] Zareba W, Moss AJ, Daubert JP, Hall WJ, Robinson JL, Andrews M. Implantable cardioverter defibrillator in high-risk long QT syndrome patients. J Cardiovasc Electrophysiol. 2003 Apr;14(4):337-41. doi: 10.1046/j.1540-8167.2003.02545.x. PMID 12741701
- [Background] Owens DK, Sanders GD, Heidenreich PA, McDonald KM, Hlatky MA. Effect of risk stratification on cost-effectiveness of the implantable cardioverter defibrillator. Am Heart J. 2002 Sep;144(3):440-8. doi: 10.1067/mhj.2002.125501. PMID 12228780
- [Background] Chatrath R, Porter CB, Ackerman MJ. Role of transvenous implantable cardioverter-defibrillators in preventing sudden cardiac death in children, adolescents, and young adults. Mayo Clin Proc. 2002 Mar;77(3):226-31. doi: 10.4065/77.3.226. PMID 11888025
- [Background] Schwartz PJ. Management of long QT syndrome. Nat Clin Pract Cardiovasc Med. 2005 Jul;2(7):346-51. doi: 10.1038/ncpcardio0239. PMID 16265560
- [Background] Quaglini S, Rognoni C, Spazzolini C, Priori SG, Mannarino S, Schwartz PJ. Cost-effectiveness of neonatal ECG screening for the long QT syndrome. Eur Heart J. 2006 Aug;27(15):1824-32. doi: 10.1093/eurheartj/ehl115. Epub 2006 Jul 13. PMID 16840497
- [Background] Yoshinaga M, Ushinohama H, Sato S, Tauchi N, Horigome H, Takahashi H, Sumitomo N, Kucho Y, Shiraishi H, Nomura Y, Shimizu W, Nagashima M. Electrocardiographic screening of 1-month-old infants for identifying prolonged QT intervals. Circ Arrhythm Electrophysiol. 2013 Oct;6(5):932-8. doi: 10.1161/CIRCEP.113.000619. Epub 2013 Sep 13. PMID 24036083
- [Background] Hayashi K, Fujino N, Uchiyama K, Ino H, Sakata K, Konno T, Masuta E, Funada A, Sakamoto Y, Tsubokawa T, Nakashima K, Liu L, Higashida H, Hiramaru Y, Shimizu M, Yamagishi M. Long QT syndrome and associated gene mutation carriers in Japanese children: results from ECG screening examinations. Clin Sci (Lond). 2009 Sep 21;117(12):415-24. doi: 10.1042/CS20080528. PMID 19371231
- [Background] Crotti L, Tester DJ, White WM, Bartos DC, Insolia R, Besana A, Kunic JD, Will ML, Velasco EJ, Bair JJ, Ghidoni A, Cetin I, Van Dyke DL, Wick MJ, Brost B, Delisle BP, Facchinetti F, George AL, Schwartz PJ, Ackerman MJ. Long QT syndrome-associated mutations in intrauterine fetal death. JAMA. 2013 Apr 10;309(14):1473-82. doi: 10.1001/jama.2013.3219. PMID 23571586
- [Background] Schwartz PJ, Stramba-Badiale M, Segantini A, Austoni P, Bosi G, Giorgetti R, Grancini F, Marni ED, Perticone F, Rosti D, Salice P. Prolongation of the QT interval and the sudden infant death syndrome. N Engl J Med. 1998 Jun 11;338(24):1709-14. doi: 10.1056/NEJM199806113382401. PMID 9624190
- [Background] Schwartz PJ. Electrocardiography first for reducing cot death. Lancet. 2001 Aug 25;358(9282):672-3. doi: 10.1016/S0140-6736(01)05809-3. No abstract available. PMID 11545089
- [Background] Hobbs JB, Peterson DR, Moss AJ, McNitt S, Zareba W, Goldenberg I, Qi M, Robinson JL, Sauer AJ, Ackerman MJ, Benhorin J, Kaufman ES, Locati EH, Napolitano C, Priori SG, Towbin JA, Vincent GM, Zhang L. Risk of aborted cardiac arrest or sudden cardiac death during adolescence in the long-QT syndrome. JAMA. 2006 Sep 13;296(10):1249-54. doi: 10.1001/jama.296.10.1249. PMID 16968849
- [Background] De Groote K, Suys B, Deleeck A, De Wolf D, Matthys D, Van Overmeire B. How accurately can QT interval be measured in newborn infants? Eur J Pediatr. 2003 Dec;162(12):875-9. doi: 10.1007/s00431-003-1321-9. Epub 2003 Oct 10. PMID 14551764
- [Background] Badilini F, Vaglio M, Sarapa N. Automatic extraction of ECG strips from continuous 12-lead holter recordings for QT analysis at prescheduled versus optimized time points. Ann Noninvasive Electrocardiol. 2009 Jan;14 Suppl 1(Suppl 1):S22-9. doi: 10.1111/j.1542-474X.2008.00260.x. PMID 19143738
- [Background] Disposable ECG electrodes. ANSI/AAMI EC12. 2000 (R2010)
- [Background] Kaltman JR, Thompson PD, Lantos J, Berul CI, Botkin J, Cohen JT, Cook NR, Corrado D, Drezner J, Frick KD, Goldman S, Hlatky M, Kannankeril PJ, Leslie L, Priori S, Saul JP, Shapiro-Mendoza CK, Siscovick D, Vetter VL, Boineau R, Burns KM, Friedman RA. Screening for sudden cardiac death in the young: report from a national heart, lung, and blood institute working group. Circulation. 2011 May 3;123(17):1911-8. doi: 10.1161/CIRCULATIONAHA.110.017228. No abstract available. PMID 21537007
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Stanley K. Design of randomized controlled trials. Circulation. 2007 Mar 6;115(9):1164-9. doi: 10.1161/CIRCULATIONAHA.105.594945. No abstract available. PMID 17339574
- [Background] Schwartz PJ, Garson A Jr, Paul T, Stramba-Badiale M, Vetter VL, Wren C; European Society of Cardiology. Guidelines for the interpretation of the neonatal electrocardiogram. A task force of the European Society of Cardiology. Eur Heart J. 2002 Sep;23(17):1329-44. doi: 10.1053/euhj.2002.3274. No abstract available. PMID 12269267
- [Background] Rautaharju PM, Surawicz B, Gettes LS, Bailey JJ, Childers R, Deal BJ, Gorgels A, Hancock EW, Josephson M, Kligfield P, Kors JA, Macfarlane P, Mason JW, Mirvis DM, Okin P, Pahlm O, van Herpen G, Wagner GS, Wellens H; American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; American College of Cardiology Foundation; Heart Rhythm Society. AHA/ACCF/HRS recommendations for the standardization and interpretation of the electrocardiogram: part IV: the ST segment, T and U waves, and the QT interval: a scientific statement from the American Heart Association Electrocardiography and Arrhythmias Committee, Council on Clinical Cardiology; the American College of Cardiology Foundation; and the Heart Rhythm Society. Endorsed by the International Society for Computerized Electrocardiology. J Am Coll Cardiol. 2009 Mar 17;53(11):982-91. doi: 10.1016/j.jacc.2008.12.014. No abstract available. PMID 19281931
- [Background] Schwartz PJ, Ackerman MJ, George AL Jr, Wilde AAM. Impact of genetics on the clinical management of channelopathies. J Am Coll Cardiol. 2013 Jul 16;62(3):169-180. doi: 10.1016/j.jacc.2013.04.044. Epub 2013 May 15. PMID 23684683
- [Background] Zou KH, O'Malley AJ, Mauri L. Receiver-operating characteristic analysis for evaluating diagnostic tests and predictive models. Circulation. 2007 Feb 6;115(5):654-7. doi: 10.1161/CIRCULATIONAHA.105.594929. No abstract available. PMID 17283280
- [Background] Newton-Cheh C, Eijgelsheim M, Rice KM, de Bakker PI, Yin X, Estrada K, Bis JC, Marciante K, Rivadeneira F, Noseworthy PA, Sotoodehnia N, Smith NL, Rotter JI, Kors JA, Witteman JC, Hofman A, Heckbert SR, O'Donnell CJ, Uitterlinden AG, Psaty BM, Lumley T, Larson MG, Stricker BH. Common variants at ten loci influence QT interval duration in the QTGEN Study. Nat Genet. 2009 Apr;41(4):399-406. doi: 10.1038/ng.364. Epub 2009 Mar 22. PMID 19305408
- [Background] Smith JG, Avery CL, Evans DS, Nalls MA, Meng YA, Smith EN, Palmer C, Tanaka T, Mehra R, Butler AM, Young T, Buxbaum SG, Kerr KF, Berenson GS, Schnabel RB, Li G, Ellinor PT, Magnani JW, Chen W, Bis JC, Curb JD, Hsueh WC, Rotter JI, Liu Y, Newman AB, Limacher MC, North KE, Reiner AP, Quibrera PM, Schork NJ, Singleton AB, Psaty BM, Soliman EZ, Solomon AJ, Srinivasan SR, Alonso A, Wallace R, Redline S, Zhang ZM, Post WS, Zonderman AB, Taylor HA, Murray SS, Ferrucci L, Arking DE, Evans MK, Fox ER, Sotoodehnia N, Heckbert SR, Whitsel EA, Newton-Cheh C; CARe and COGENT consortia. Impact of ancestry and common genetic variants on QT interval in African Americans. Circ Cardiovasc Genet. 2012 Dec;5(6):647-55. doi: 10.1161/CIRCGENETICS.112.962787. Epub 2012 Nov 19. PMID 23166209
- [Background] Seeb JE, Pascal CE, Ramakrishnan R, Seeb LW. SNP genotyping by the 5'-nuclease reaction: advances in high-throughput genotyping with nonmodel organisms. Methods Mol Biol. 2009;578:277-92. doi: 10.1007/978-1-60327-411-1_18. PMID 19768601
- [Background] Shen GQ, Abdullah KG, Wang QK. The TaqMan method for SNP genotyping. Methods Mol Biol. 2009;578:293-306. doi: 10.1007/978-1-60327-411-1_19. PMID 19768602
- [Background] Pearl W. Effects of gender, age, and heart rate on QT intervals in children. Pediatr Cardiol. 1996 May-Jun;17(3):135-6. doi: 10.1007/BF02505201. PMID 8662028
- [Background] Zhang Y, Post WS, Dalal D, Blasco-Colmenares E, Tomaselli GF, Guallar E. Coffee, alcohol, smoking, physical activity and QT interval duration: results from the Third National Health and Nutrition Examination Survey. PLoS One. 2011 Feb 28;6(2):e17584. doi: 10.1371/journal.pone.0017584. PMID 21386989
- [Background] Huang H, Amin V, Gurin M, Wan E, Thorp E, Homma S, Morrow JP. Diet-induced obesity causes long QT and reduces transcription of voltage-gated potassium channels. J Mol Cell Cardiol. 2013 Jun;59:151-8. doi: 10.1016/j.yjmcc.2013.03.007. Epub 2013 Mar 19. PMID 23517696
- [Background] Howard PA. Azithromycin-induced proarrhythmia and cardiovascular death. Ann Pharmacother. 2013 Nov;47(11):1547-51. doi: 10.1177/1060028013504905. PMID 24285766
- [Background] Katz DF, Sun J, Khatri V, Kao D, Bucher-Bartelson B, Traut C, Lundin-Martinez J, Goodman M, Mehler PS, Krantz MJ. QTc interval screening in an opioid treatment program. Am J Cardiol. 2013 Oct 1;112(7):1013-8. doi: 10.1016/j.amjcard.2013.05.037. Epub 2013 Jun 29. PMID 23820570
- [Background] Villain E, Levy M, Kachaner J, Garson A Jr. Prolonged QT interval in neonates: benign, transient, or prolonged risk of sudden death. Am Heart J. 1992 Jul;124(1):194-7. doi: 10.1016/0002-8703(92)90940-w. PMID 1352080
- [Background] Arking DE, Pulit SL, Crotti L, van der Harst P, Munroe PB, Koopmann TT, Sotoodehnia N, Rossin EJ, Morley M, Wang X, Johnson AD, Lundby A, Gudbjartsson DF, Noseworthy PA, Eijgelsheim M, Bradford Y, Tarasov KV, Dorr M, Muller-Nurasyid M, Lahtinen AM, Nolte IM, Smith AV, Bis JC, Isaacs A, Newhouse SJ, Evans DS, Post WS, Waggott D, Lyytikainen LP, Hicks AA, Eisele L, Ellinghaus D, Hayward C, Navarro P, Ulivi S, Tanaka T, Tester DJ, Chatel S, Gustafsson S, Kumari M, Morris RW, Naluai AT, Padmanabhan S, Kluttig A, Strohmer B, Panayiotou AG, Torres M, Knoflach M, Hubacek JA, Slowikowski K, Raychaudhuri S, Kumar RD, Harris TB, Launer LJ, Shuldiner AR, Alonso A, Bader JS, Ehret G, Huang H, Kao WH, Strait JB, Macfarlane PW, Brown M, Caulfield MJ, Samani NJ, Kronenberg F, Willeit J; CARe Consortium; COGENT Consortium; Smith JG, Greiser KH, Meyer Zu Schwabedissen H, Werdan K, Carella M, Zelante L, Heckbert SR, Psaty BM, Rotter JI, Kolcic I, Polasek O, Wright AF, Griffin M, Daly MJ; DCCT/EDIC; Arnar DO, Holm H, Thorsteinsdottir U; eMERGE Consortium; Denny JC, Roden DM, Zuvich RL, Emilsson V, Plump AS, Larson MG, O'Donnell CJ, Yin X, Bobbo M, D'Adamo AP, Iorio A, Sinagra G, Carracedo A, Cummings SR, Nalls MA, Jula A, Kontula KK, Marjamaa A, Oikarinen L, Perola M, Porthan K, Erbel R, Hoffmann P, Jockel KH, Kalsch H, Nothen MM; HRGEN Consortium; den Hoed M, Loos RJ, Thelle DS, Gieger C, Meitinger T, Perz S, Peters A, Prucha H, Sinner MF, Waldenberger M, de Boer RA, Franke L, van der Vleuten PA, Beckmann BM, Martens E, Bardai A, Hofman N, Wilde AA, Behr ER, Dalageorgou C, Giudicessi JR, Medeiros-Domingo A, Barc J, Kyndt F, Probst V, Ghidoni A, Insolia R, Hamilton RM, Scherer SW, Brandimarto J, Margulies K, Moravec CE, del Greco M F, Fuchsberger C, O'Connell JR, Lee WK, Watt GC, Campbell H, Wild SH, El Mokhtari NE, Frey N, Asselbergs FW, Mateo Leach I, Navis G, van den Berg MP, van Veldhuisen DJ, Kellis M, Krijthe BP, Franco OH, Hofman A, Kors JA, Uitterlinden AG, Witteman JC, Kedenko L, Lamina C, Oostra BA, Abecasis GR, Lakatta EG, Mulas A, Orru M, Schlessinger D, Uda M, Markus MR, Volker U, Snieder H, Spector TD, Arnlov J, Lind L, Sundstrom J, Syvanen AC, Kivimaki M, Kahonen M, Mononen N, Raitakari OT, Viikari JS, Adamkova V, Kiechl S, Brion M, Nicolaides AN, Paulweber B, Haerting J, Dominiczak AF, Nyberg F, Whincup PH, Hingorani AD, Schott JJ, Bezzina CR, Ingelsson E, Ferrucci L, Gasparini P, Wilson JF, Rudan I, Franke A, Muhleisen TW, Pramstaller PP, Lehtimaki TJ, Paterson AD, Parsa A, Liu Y, van Duijn CM, Siscovick DS, Gudnason V, Jamshidi Y, Salomaa V, Felix SB, Sanna S, Ritchie MD, Stricker BH, Stefansson K, Boyer LA, Cappola TP, Olsen JV, Lage K, Schwartz PJ, Kaab S, Chakravarti A, Ackerman MJ, Pfeufer A, de Bakker PI, Newton-Cheh C. Genetic association study of QT interval highlights role for calcium signaling pathways in myocardial repolarization. Nat Genet. 2014 Aug;46(8):826-36. doi: 10.1038/ng.3014. Epub 2014 Jun 22. PMID 24952745
- [Background] Saul JP, Schwartz PJ, Ackerman MJ, Triedman JK. Rationale and objectives for ECG screening in infancy. Heart Rhythm. 2014 Dec;11(12):2316-21. doi: 10.1016/j.hrthm.2014.09.047. Epub 2014 Sep 18. PMID 25239430
- [Background] Skinner JR, Van Hare GF. Routine ECG screening in infancy and early childhood should not be performed. Heart Rhythm. 2014 Dec;11(12):2322-7. doi: 10.1016/j.hrthm.2014.09.046. Epub 2014 Sep 18. PMID 25239431
- [Background] Saul JP, Schwartz PJ, Ackerman MJ, Triedman JK. Neonatal ECG screening: opinions and facts. Heart Rhythm. 2015 Mar;12(3):610-611. doi: 10.1016/j.hrthm.2014.11.032. Epub 2014 Dec 10. No abstract available. PMID 25499628